CLINICAL TRIAL: NCT04185194
Title: Effect of Lidocaine Phonophoresis Versus Pulsed Ultrasound on Myofascial Pain Syndrome in Athletic Children
Acronym: PH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed abdel Moneim Abo El Roos, pediatric physical therapy specialist (master degree), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/001708
Record Dates: First submitted 2019-11-15; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Treatment Side Effects
Keywords: myofascial pain syndrome, pain quality
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Participant
Masking Description: sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group A (Active Comparator): received especially designed physical therapy program
  Interventions: Other: especially designed physical therapy program
- group b (Experimental): received pulsed ultrasound in addition to physical therapy program
  Interventions: Drug: Lidocaine; Device: pulsed ultrasound; Other: especially designed physical therapy program
- group c (Experimental): received lidocaine phonophoresis in addition to physical therapy program
  Interventions: Drug: Lidocaine; Device: pulsed ultrasound; Other: especially designed physical therapy program

INTERVENTIONS:
Drug: Lidocaine — transmission of the drug molecules to the underlying muscles
  Other Names: lidocaine topical
  Arms: group b; group c
Device: pulsed ultrasound — using thermogenic and cavitation effect of ultrasound to reduce tight muscles and relieve pain
  Arms: group b; group c
Other: especially designed physical therapy program — by myofascial trigger point release, stretching and strengthening exercises of upper trapezius muscle and infrared radiation by tungsten lamp for upper trapezius

SUMMARY:
A topical anesthetic gel lidocaine has been widely used as a local anesthetic to reduce the pain and discomfort. It provides local analgesia by blocking the initiation and transmission of impulses. Lidocaine topical anesthetic gel allows the use of high concentrations of the anesthetic bases without concern about local irritation, uneven absorption or systemic toxicity (Argoff, 2000 ). So, the aim of this study is to compare between the effect of lidocaine phonophoresis and pulsed ultrasound in myofascial pain syndrome in swimmers children.

DETAILED DESCRIPTION:
Fourty five children (athletic swimmers) participated in this study, and were classified into three groups ; First control group A : this group consisted of fifteen children were receiving traditional physical therapy program. Second study group B: this group consisted of fifteen children were receiving pulsed ultrasound in addition to traditional physical therapy program as the same as in group A. Third study group C: this group consisted of fifteen children were receiving lidocaine phonophoresis in addition to traditional physical therapy program as the same as in group A. Treatment program in the three groups applied three times a week for three successive months. The study was done in the outpatient clinic of Ismailiy Sporting Club, Ismailia, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* • Age range from 10 to 14 years.

  * All children have regional neck pain complaint.
  * Tenderness in cervical trigger points in the midpoint of the upper border of trapezius muscle, from grade II to grade IV according to tenderness grading scheme (Hubbard and Berkoff, 1993) (Appendix I ) ● The diagnosis of an active MTrP in the upper trapezius according to (Ardiçet al . , 2002 and Bruno, 2005)

Exclusion Criteria:

* • Neurological disorders.

  * Dermatological disorders.
  * Acute trauma prior to the study.
  * Fibromyalgia, systemic disease and drug allergy history were excluded from the study.
  * Having myofascial trigger points injection.
  * Chronic pain in both sides of the body.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
interleukin 6 | three months
  measurement of interleukin 6 cncentration in blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Asser Sallam, PhD, Study Director — Suez Canal University
Locations (1):
- faculty of physical therapy,Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
results of the study design, abstract, conclusion